| 1 | |
|---|---|
| 2 | |
| 3 | |
| 4 | |
| 5 | Title: Randomized Controlled Trial Comparing Clinical and Radiological Outcomes |
| 6 | Between C3 Laminectomy with C4-C6 Laminoplasty and C3-C6 Laminoplasty |
| 7 | |
| 8 | Study protocol (date: 2017-01-05) |
| 9 | |

## Background

- 2 C3 laminectomy in cervical laminoplasty is a modified laminoplasty technique that can
- 3 preserve semispinalis cervicis muscle attached to the C2 spinous process. Several previous
- 4 studies have shown that this technique can lead to better outcomes of postoperative axial neck
- 5 pain and C2-C3 range of motion (ROM) than conventional cervical laminoplasty. However,
- 6 there is still a lack of understanding of total and proportional postoperative cervical sagittal
- 7 alignment outcomes.

8

9

1

## Study design

- A randomized clinical trial will be conducted on patients with cervical laminoplasty for
- treating CSM or OPLL at a single tertiary referral university hospital. Patients will be
- randomly assigned to either the LN group (C4-6 laminoplasty with C3 laminectomy) or the
- LP group (C3-6 laminoplasty) at a 1:1 ratio. The sample size will be calculated to achieve a
- target of 80% power with a two-tailed significance level of 0.05, with a medium effect size
- (Cohen's d = 0.50), resulting in 63 patients per each group. The trial will enrolled consecutive
- patients who underwent cervical laminoplasty from March 2017. Participants' ages will
- ranged from 20 to 80 years. Patients with metastatic tumors, combined fractures, or previous
- posterior cervical surgeries will be excluded from this study. Patients with a diagnosis of
- 19 CSM or OPLL will be assessed prior to randomization by a neurosurgical specialist through a
- 20 combination of history-taking, clinical examination, and radiological workup, including
- 21 dynamic radiographs and cervical spine computer tomography (CT) or magnetic resonance
- image (MRI) scans. Diagnosis of CSM will be based on symptoms of myelopathy and
- stenosis at two or more cervical levels on MRI. Diagnosis of OPLL will be made based on
- 24 CT findings. The randomization process, surgical group options, and required follow-up
- evaluations and imaging will be fully explained to eligible patients by a neurosurgical

- specialist. After obtaining informed consent, patients will be randomized using a computer-
- 2 generated block design in 1:1 ratio with concealed assignment managed by an independent
- 3 research nurse. The attending surgeons, patients, and staff members in the operating room
- 4 will be blinded to the surgical method until the day of surgery. A concealed paper indicating
- 5 the patient's assigned group will be provided in the operating room, and the surgeon will
- 6 verify the patient's group just before commencing the surgery. This study was approved by
- 7 the hospital's Institutional Review Board (IRB number: H-1610-136-804).

8

9

## **Data collection and outcomes**

- Data will be collected using patient-reported outcome questionnaires and plain x-rays taken at
- the outpatient clinic before surgery and at 1, 2, and 3 years postoperatively. Patients will
- record their outcomes directly without assistance of the surgeon or other study participants.
- Radiological parameters will be assessed using 150% magnified images by one of the authors
- 14 (a fellow). Three measurements will be performed, and the median value will be selected as
- the final measurement. The measurements will be conducted utilizing the measuring tools
- within the institution's Picture Archiving and Communication System (M6, Infinitt
- Healthcare, Seoul, Korea) operating on a Microsoft Windows environment (Microsoft Corp.,
- 18 Redmond, WA, USA). We selected C2-C7 Cobb angle (C2-C7 CA) as the primary outcome
- measure, considering the importance of postoperative kyphotic changes in cervical
- laminoplasty, which have been associated with long-term recurrent myelopathy and chronic
- 21 neck pain. Additionally, we chose the Neck Disability Index (NDI) as another primary
- outcome measure to evaluate axial neck pain, as it is commonly acknowledged as a potential
- 23 advantage of C3 laminectomy. Secondary outcome measures included other radiologic
- parameters such as C2-C3 Cobb angle (C2-C3 CA), C4-C7 Cobb angle (C4-C7 CA), cervical
- sagittal vertical axis (cSVA), T1 slope (T1S) and T1 slope minus cervical lordosis (T1S-CL),

- as well as presence of C2-C3 interlaminar fusion. Other clinical outcomes, such as numerical
- 2 rating scores for neck (NRS-N) and limb (NRS-L) and the Euro-Quality of Life-5 Dimension
- 3 (EQ-5D), will be also assessed. We will examine operation-related factors, including open
- 4 side, presence of dome-like laminectomy at the C2 or C7 level, operative time, estimated
- 5 blood loss, and complications such as hinge fracture, neural injury, dural injury, and wound
- 6 infection.

7

8

## Statistical analysis plan

- 9 Outcomes will be analyzed using the modified intention-to-treat (mITT) strategy. The mITT
- population will consist of all participants with randomly assigned surgery and have available
- at least a year of postoperative data from 1 to 3 years. Baseline and operation-related
- characteristics of the LN and LP groups will be compared using independent t-tests for
- continuous variables, and chi-square tests or Fisher's exact tests for categorical variables.
- Postoperative clinical outcomes and radiological parameters will be compared between
- groups and over time using linear mixed-effects models, with fixed effects including
- preoperative values of tested variables, group, time, interaction between group and time,
- other factors with possible relation with outcomes such as age, BMI and disease, and a
- random effect of subjects. Least squares mean for postoperative clinical outcomes and
- radiological parameters will be estimated. Comparisons will be made between the treatment
- 20 groups. For variables with a significant difference in the interaction between time and group,
- 21 post-hoc analysis will be performed for each time point and adjusted p-values will be
- evaluated using the Bonferroni method. All data will be analyzed using SPSS software
- version 27.0 (SPSS, Chicago, IL, USA), with statistical significance defined at p < 0.05 (two-
- 24 sided).